CLINICAL TRIAL: NCT03957980
Title: Remote Access to Care for Children With Cortical Visual Impairment and Their Families
Brief Title: Remote Access: Cortical Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0356
Record Dates: First submitted 2019-05-03; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Cortical Visual Impairment
MeSH Terms: conditions — Blindness, Cortical | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This pilot study will utilize a randomized two group crossover design with assessment at 4 time periods.
Who Masked: Outcomes Assessor
Masking Description: The occupational therapist at the remote clinics assessing outcomes did not know what point in time the subjects were receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention First (Other): The participants in this arm of the study received occupational therapy via telehealth in the first 12 weeks of enrollment, then received no other intervention for the duration of the study.
  Interventions: Other: Occupational therapy
- No Intervention First (Other): The participants in this arm of the study did not receive an intervention in the first 12 weeks of enrollment, but received occupational therapy via telehealth during the second 12 weeks of enrollment.
  Interventions: Other: Occupational therapy

INTERVENTIONS:
Other: Occupational therapy — Child/caregiver dyads in this group will participate in telehealth-based intervention sessions in their home environment. Each child/caregiver dyad will participate in up to 9 interventions sessions. All intervention sessions will last 30-60 minutes. The intervention sessions will focus on task analysis, caregiver coaching, parent education and recommendations for task and home/environmental modifications to promote the child's functional vision.

SUMMARY:
This study aims to compare the efficacy of an in-home telehealth-based intervention to standard care for children with cortical visual impairment and their caregivers and to assess the feasibility and acceptability of an in-home telehealth-based intervention approach for children with cortical visual impairment and their caregivers. This pilot study will utilize a randomized two group crossover design with assessment at 4 time periods. The assessments will occur at remote locations.

DETAILED DESCRIPTION:
To improve access to evaluation and treatment, the investigators will be offering remote cortical visual impairment clinics to assess children for cortical visual impairment. The cortical visual impairment clinics will be organized in public spaces such as school buildings, libraries, and/or hospital clinics. Study staff will contact potential clinics, buildings, etc., about interest in hosting these remote clinics. The cortical visual impairment clinics will be staffed by at least one of the following individuals: an ophthalmologist and/or an optometrist, a technician, and an occupational therapist. All participants will attend 4 remote cortical visual impairment clinics during the study. Prior to the initial clinic visit, the participants will be randomized into either the waitlist control group or the intervention group using the list of patients scheduled for the clinic. During the initial clinic visit, each child who has been given parental consent will complete both an eye exam (either an ophthalmologist or an optometrist) and functional vision evaluation with an occupational therapist. Both the eye exam and the functional vision evaluation occurring during the clinic visit are the same as would be provided during routine clinical care. None of the examinations provided during this research study will be billed through insurance. Those who are diagnosed with cortical visual impairment will continue on with the study. The intervention group will complete the telehealth intervention sessions and the waitlist control group will continue with standard care. All participants will attend three additional cortical visual impairment Clinics: one 4 months after the initial evaluation (+/- 2 weeks), one 8 months after initial evaluation (+/- 2 weeks) and another 12 months after the initial evaluation (+/- 2 weeks). During the final three cortical visual impairment clinics, the participants will complete and updated Cortical Visual Impairment Range and Canadian Occupational Performance Measure with the occupational therapist.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 months to 6 years 11 months with suspected or previously diagnosed Cortical Visual Impairment If the child has previously diagnosed Cortical Visual Impairment, they receive regular ongoing therapy related to vision, no more than one time/session a week at the time of recruitment.
* Caregivers of the children with suspected/ diagnosed Cortical Visual Impairment need to be cognitively able to provide meaningful consent and parent permission in order to be included in the study
* Home address must be in either Ohio, Kentucky, West Virginia or Indiana (due to Occupational Therapy licensure laws and telehealth).
* English speaking

Exclusion Criteria:

* Children who were not referred for an evaluation for Cortical Visual Impairment
* Children who don't live in Ohio, Kentucky, Indiana, or West Virginia
* Children who are already receiving more than one therapy sessions related to vision a week

Ages: 12 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Change in Functional Vision as measured by the Cortical Visual Impairment Range | Collected at the Initial Remote Clinic and the 4-month follow up clinic for the intervention first group and the 8-month follow up clinic for the no intervention first group
  the Cortical Visual Impairment Range is a reliable assessment utilized to measure functional vision for children with Cortical Visual Impairment.. The Cortical Visual Impairment Range consists of 10 behavioral characteristics common in children with Cortical Visual Impairment. Each behavioral characteristic is rated on a scale from 0-1. The characteristic scores are summed to get an overall score of functional vision. This score will be treated as a continuous variable for analysis.

SECONDARY OUTCOMES:
Change in Individualized, function goals as measured by the Canadian Occupational Performance Measure (COPM) | The COPM will be completed before the intervention, at month 4 in clinic, month 8 (via phone/ email/ mail) and month 12 in clinic (all +/- 2 weeks).
  The COPM is a valid, reliable, and responsive assessment tool (28-30) that measures the caregiver's perception of the child's performance on goals that are important to the child and his/her caregiver. The COPM will help guide the treatment plan for the Cortical Visual Impairment interventions. Overall satisfaction and performance scores are generated from the COPM and each will be treated as a continuous variable for analysis.
Change in Individualized, function goals as measured by the Preverbal Visual Assessment (PreVias) | The PreVias will be completed before the intervention, at month 4 in clinic, month 8 (via phone/ email/ mail) and month 12 in clinic (all +/- 2 weeks).
  The PreVias is a questionnaire to be completed by the caregiver. It has 30 questions related to one or more visual domain including visual attention, visual communication, visual-motor coordination and visual processing.

OTHER OUTCOMES:
Caregiver and Therapist Telehealth Qualitative Data | Completed at the end of the Initial Remote Clinic visit (consent is obtained and an eye exam is completed here; the survey is filled out immediately following the eye exam)
  A questionnaire will be given to both the intervention and control group. This survey asks questions regarding the quality and the quantity of information given at the initial evaluation. The survey is in a multiple choice format and the answer options range from Strongly Disagree to Strongly Agree (Strongly Agree indicates a positive response.
Caregiver and Therapist Intervention Questionnaire | Completed at the 4-month Follow Up Remote Clinic for the Intervention First group and completed at the 8-month Follow Up Remote Clinic for the No Intervention First group
  The questionnaire will gather data regarding how the therapist and caregiver felt regarding the number of sessions, the set up, the child's improvement, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available to other researchers.